CLINICAL TRIAL: NCT00312572
Title: A Randomized, Double-Blind Study Evaluating the Dose Conversion From Vicodin® to Buprenorphine Transdermal System (BTDS) in Subjects With Osteoarthritis (OA) Pain
Brief Title: Safety and Efficacy of Dose Conversion From Vicodin® to Buprenorphine Transdermal System (Butrans™) in Subjects With OA Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BUP3018
Record Dates: First submitted 2006-04-07; First posted 2006-04-10 (Estimated); Results first posted 2010-09-23 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis, opioid, transdermal
MeSH Terms: conditions — Osteoarthritis | interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- BTDS10/20 (Experimental): Initial doses (Level 1) of BTDS 10. Subjects were allowed to have their doses adjusted to BTDS 20 (Level 2) on or after day 4.
  Interventions: Drug: Buprenorphine transdermal patch
- BTDS 20 (Experimental): Initial doses (Level 1) of BTDS 20.
  Interventions: Drug: Buprenorphine transdermal patch

INTERVENTIONS:
Drug: Buprenorphine transdermal patch — Buprenorphine transdermal patch applied for 7-day wear.
  Other Names: Butrans™

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of dose conversion from hydrocodone/ acetaminophen (Vicodin®) to the buprenorphine transdermal system (Butrans™) in subjects with osteoarthritis pain of the hip or knee. The double-blind treatment intervention duration is 2 weeks during which time supplemental analgesic medication will be allowed.

DETAILED DESCRIPTION:
Buprenorphine is a synthetic opioid analgesic with over 25 years of international clinical experience indicating it to be safe and effective in a variety of therapeutic situations for the relief of moderate to severe pain.

ELIGIBILITY:
Inclusion Criteria:

- osteoarthritis of the hip or knee taking a regularly scheduled regimen of hydrocodone/ acetaminophen for their osteoarthritis OA pain.

Exclusion Criteria:

* currently have condition requiring a stable regimen of acetaminophen (APAP).
* a history of chronic conditions, other than OA of the hip or knee joints, requiring frequent, intermittent analgesic therapy.

Other protocol-specific exclusion/inclusion criteria may apply.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2003-06; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- United States (36):
  - Southern Drug Research, Birmingham, Alabama
  - Redpoint Research, Phoenix, Arizona
  - Advanced Clinical Therapeutics, Tucson, Arizona
  - Tucson Orthopedic Institute, Tucson, Arizona
  - Hot Springs Mercy Pain Clinic, Hot Springs, Arkansas
  - Private Practice, Pine Bluff, Arkansas
  - Advanced Clinical Research Institute, Anaheim, California
  - Lovelace Scientific Resources, Beverly Hills, California
  - Southbay Pharma Research, Buena Park, California
  - Community Medical Providers, Clovis, California
  - Kaiser Permanente, Escondido, California
  - Univ. of Southern California, Santa Monica, California
  - Arthritis Center of CT, Waterbury, Connecticut
  - Lifespan Research Foundation, Inc., Miami, Florida
  - Miami Beach Anesthesiology Associates, Miami Beach, Florida
  - Neuro Science and Spine Assoc., Naples, Florida
  - West Broward Rheumatology Association, Inc., Tamarac, Florida
  - Intermountain Orthopaedics, Boise, Idaho
  - University of Kansas Medical Center, Kansas City, Kansas
  - Bluegrass Orthopaedics, Lexington, Kentucky
  - Commonwealth Biomedical Research, LLC, Madisonville, Kentucky
  - Dolby Providers, Inc., New Orleans, Louisiana
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Westside Family Medical Center, Kalamazoo, Michigan
  - PCM Medical Services, Lansing, Michigan
  - HealthCare Research LLC, St Louis, Missouri
  - Northeast Pain Research Center, Barrington, New Hampshire
  - The Arthritis Clinic and Carolina Bone and Joint, Charlotte, North Carolina
  - Dayton Primary and Urgent Care, Dayton, Ohio
  - The Medford Medical Clinic, Medford, Oregon
  - The Arthritis and Osteoporosis Center, Orangeburg, South Carolina
  - CEDRA Clinical Research,, Austin, Texas
  - Renaissance Clinical Research & Hypertension Clinic, Dallas, Texas
  - Spine Care Southwest., Houston, Texas
  - KRK Medical Research, Richardson, Texas
  - Monroe Medical Foundation, Monroe, Wisconsin

REFERENCES:
- [Result] Ripa SR, McCarberg BH, Munera C, Wen W, Landau CJ. A randomized, 14-day, double-blind study evaluating conversion from hydrocodone/acetaminophen (Vicodin) to buprenorphine transdermal system 10 mug/h or 20 mug/h in patients with osteoarthritis pain. Expert Opin Pharmacother. 2012 Jun;13(9):1229-41. doi: 10.1517/14656566.2012.667073. Epub 2012 Mar 12. PMID 22409388

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study dates: 26-Jun-2003 (first patient first visit) to 21-Jul-2004 (last patient last visit) in 29 medical/research centers in the United States.
Pre-assignment Details: N = 266 subjects received a stable regimen of Vicodin® in the Run-in period and were eligible for randomization if they reported a daily "average pain over the last 24 hours" score of 0=none or 1=mild on at least 5 of the 7 days; and used ≤ 2 doses of supplemental analgesic per day for their osteoarthritic (OA) pain. N = 204 completed the run-in.
Groups:
- Double-blind BTDS 10/20: Initial doses (Level 1) of BTDS 10. Subjects were allowed to have their dose adjusted to BTDS 20 (Level 2) on or after day 4. Subjects remained on their treatment regimen until day 14 (± 2 days) or until they discontinued from the study. Downward titration was not permitted.
- Double-blind BTDS 20: Initial doses (Level 1) of BTDS 20. Subjects remained on their treatment regimen until day 14 (± 2 days) or until they discontinued from the study. Downward titration was not permitted.
Period: Overall Study
Arm/Group | Double-blind BTDS 10/20 | Double-blind BTDS 20
Started | 101 | 103
Completed | 85 | 82
Not Completed | 16 | 21
Not completed — Adverse Event | 10 | 16
Not completed — Lost to Follow-up | 1 | 1
Not completed — Administrative | 4 | 2
Not completed — Lack of Efficacy | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-blind BTDS 10/20 | Double-blind BTDS 20 | Total
Number analyzed (Participants) | 101 | 103 | 204
Age Continuous [Mean (Standard Deviation); unit: years] | 57.4 (10.10) | 58.9 (9.97) | 58.2 (10.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 73 | 136
  Male | 38 | 30 | 68

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects Who Completed the 14-day Double-blind Phase.
Description: The indicator variable was 1 = completion, and 0 = noncompletion. For the primary efficacy analysis, the percentage of subjects who completed the double-blind phase was computed with its 95% confidence interval (CI) for each treatment regimen (starting dose of BTDS 10 or BTDS 20) across and within baseline Vicodin® stratum (15 to 22.5mg/day vs >22.5 to 30 mg/day as determined by the daily average hydrocodone dose during the run-in period).
Time Frame: 14 days
Population: Full Analysis Population: (N = 198) consisted of all subjects who were randomized into the double-blind phase, received at least 1 dose of BTDS during the double-blind phase, and had at least 1 efficacy observation during the double-blind phase, and had no evidence of impaired liver function at screening and prerandomization.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Combined Total: Combined percentages from BTDS 10/20 and BTDS 20
Arm/Group | Double-blind BTDS 10/20 | Double-blind BTDS 20 | Combined Total
Number analyzed (Participants) | 98 | 100 | 198
Percentage of Participants
  15 - 22.5 mg HCD (Stratum 1) | 88 [79.9 to 95.1] | 83 [74.7 to 91.9] | 85 [79.7 to 91.2]
  more than 22.5 - 30 mg HCD (Stratum 2) | 85 [70.8 to 98.5] | 79 [63.4 to 93.8] | 82 [71.1 to 91.8]
  Overall | 87 [80.0 to 93.5] | 82 [74.5 to 89.5] | 84 [79.3 to 89.4]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) that occurred after the signing of the informed consent up to end of study and followed until resolution or 30 days after the last dose of study drug, or discontinuation; serious AEs were followed until the AE stabilized
Description: AEs were learned of through spontaneous reports and subject interview.
Groups:
- Open-label Run-in Period - Vicodin: N = 266 subjects received a stable regimen of Vicodin® in the Run-in period and were eligible for randomization if they reported a daily "average pain over the last 24 hours" score of 0 = none or 1 = mild on at least 5 of the 7 days; and used ≤ 2 doses of supplemental analgesic per day for their osteoarthritic (OA) pain. N = 204 completed the run-in.
Arm/Group | Double-blind BTDS 10/20 | Double-blind BTDS 20 | Open-label Run-in Period - Vicodin
Serious Adverse Events (participants affected / at risk) | 2/101 | 3/103 | 0/266
Other Adverse Events (participants affected / at risk) | 31/101 | 47/103 | 15/266
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind BTDS 10/20 (N=101) | Double-blind BTDS 20 (N=103) | Open-label Run-in Period - Vicodin (N=266)
Creutzfeldt-Jacob disease - DEATH (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — DEATH Systematic and nonsystematic assessments
Exacerbation of anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessments
Increased hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessments
Leg pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessments
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessments
Rash NOS, Chest, Arms, Face (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments
Rash generalized (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments
OTHER ADVERSE EVENTS (reported when occurring in more than 4.50% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind BTDS 10/20 (N=101) | Double-blind BTDS 20 (N=103) | Open-label Run-in Period - Vicodin (N=266)
Application site erythema (General disorders) | 7 | 7 | 0
Application site pruritus (General disorders) | 11 | 18 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 8 | 0
Dizziness (Nervous system disorders) | 3 | 7 | 1
Headache (Nervous system disorders) | 9 | 9 | 6
Nausea (Gastrointestinal disorders) | 10 | 10 | 4
Somnolence (Nervous system disorders) | 7 | 9 | 1
Vomiting NOS (Gastrointestinal disorders) | 6 | 7 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days